CLINICAL TRIAL: NCT06499506
Title: Skew Flap vs Long Posterior Flap for Below Knee Amputation Early and Short- Term Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Abdelmageed, Ibrahim, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-06-15MS
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot; Ischemic Leg
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: comparison between Skew flap and long posterior flap for below knee amputation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skew Flap (Active Comparator): skew Flap technique for below knee amputation
  Interventions: Procedure: Below knee amputation
- Long Posterior Flap (Active Comparator): Long Posterior Flap for Below knee amputation
  Interventions: Procedure: Below knee amputation

INTERVENTIONS:
Procedure: Below knee amputation — trans tibial amputation one hand breadth below tibial tuberosity

SUMMARY:
Below knee amputations (BKAs) are frequently performed among vascular patients with end stage chronic limb threatening ischemia and / or complications of diabetes and diabetic foot infections and gangrene, It may also be necessary for patients with aggressive diabetic foot infections or gangrene, or both; for those with extensive venous ulceration; or following major trauma. and in the case of extremity sepsis.

There is two main methods for constructing the myocutaneous flaps in below knee amputation; the long posterior flap (LPF) and skew flap (SF).

DETAILED DESCRIPTION:
Anesthesia BKA could be performed under general anesthesia (GA), epidural anesthesia or under spinal anesthesia .

Patient position The patient lies in the supine position. Technique The limb is prepared by an application of povidone iodine solution in the ward 2 h before surgery. The foot and any septic lesion is isolated. The whole limb is wrapped in a dry sterile sheet. Penicillin and metronidazole prophylaxis is used routinely.

The operation is performed under general anesthesia with a regional anesthetic technique.

The skin flaps are marked on the skin before any incision. And the skin flaps are semicircular. based on a line around the limb at right angles to its long axis, drawn at the plane of bone section 10-12cm from the joint line at the tibial plateau.

The skin flaps are cut which includes the fat and deep fascia. but these are not stripped from the underlying muscle more than is required to gain access to the anterior tibial compartment. The saphenous veins are ligated. The periosteum over the tibia is incised where it is exposed and elevated with the skin flap to 2 cm above the line of bone section.

The anterior tibial nerve and the peroneal nerve are divided and allowed to retract while the vessels are ligated. The fibula is divided 2cm above the line of tibial bone section.

The tibia is divided with a GIGLI saw. Traction on the bone hook exposes the tibialis posterior muscle and this is divided at the line of distal bone section which exposes the posterior tibial artery and its venae comitantes. the posterior tibial nerve and the peroneal artery and its venae comitantes. ligatures applied to each of the vascular bundles. The gastrocnemius and soleus muscle mass can then be separated from the tibia and fibula of the specimen while hemostasis is maintained. The muscle mass is cut transversely, thus freeing the specimen; this must allow a length of muscle below the bone end at least equal to the diameter of the leg.

The protruding muscle mass is then thinned from the line of bone section to its extremity .

Careful homeostasis is essential and the muscle must not be compressed due to too much bulk or tight constricting sutures.

A suction tube drain is drawn through the lateral aspect of the stump above the suture line and placed to collect any fluid in the vicinity of the bone ends.

The drain can be removed in 48-72 h; the sutures are removed at 15- 21 days. Follow up Patients will be followed up prospectively intraoperative, during postoperative hospital admission and late in outpatient clinic.

Major adverse clinical events (MACE) are carefully monitored. Follow up include immediate postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic atherosclerotic occlusive disease of the lower extremity and threatening limb ischemia (intractable rest pain, ulcer or gangrene) for whom all other treatment options failed or inapplicable .
* patients with aggressive diabetic foot infections or gangrene, or both.
* Patients with extensive venous ulceration.
* Patients following major trauma with unsalvageable limb.
* Patients with nonfunctioning damaged limb as in Charcot joint disease.
* Patients with extensive limb sepsis.

Exclusion Criteria:

* Patients with local site infection not candidate for instant closure.
* Patients with bad general condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Healing | 6 month
  Primary stump healing, defined as a painless, healed suture line enabling fitting of a prosthetic limb (if appropriate) and regaining of mobility
Re ampuation | 1 month
  Rate of reamputation at (a) same level; (b) higher level.
Mobilization | 6 month
  Number of participants mobilizing with a prosthetic limb.

SECONDARY OUTCOMES:
Mortality | 1 month
  Thirty-day mortality rate.
Hospital stay | 1 month
  Length of hospital stay.
complaints | 2 month
  Symptoms relating to the stump, such as pain and swelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided